CLINICAL TRIAL: NCT05927090
Title: Surgical Strategy for Repair of Aortic Dissection: A Multicenter Registry
Brief Title: Outcomes of Aortic Dissection Repair
Acronym: STAAD
Status: Enrolling by invitation | Type: Observational
Sponsor: Centre Cardiologique du Nord (Other)
Collaborators: Henri Mondor University Hospital (Other); Universita degli Studi di Genova (Other); Pitié-Salpêtrière Hospital (Other); Ospedale San Camillo, Rome, Italy (Unknown); Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Francesco Nappi, Doctor, Centre Cardiologique du Nord
Other Study IDs: CN-202201173-3; CN-202201173-3 (Registry Identifier: STAD-Registry)
Record Dates: First submitted 2023-06-03; First posted 2023-07-03 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Type A Aortic Dissection; Ascending Aortic Dissection; Aortic Diseases; Aortic Arch; Aortic Valve Insufficiency; Aortic Root Dissection; Aortic Root Dilatation; Type B Aortic Dissection
Keywords: DeBakey type I Dissection; DeBakey type II Dissection; Type A Acute Aortic Dissection (TAAAD); Root-Sparing Replacement; Ascending Aorta Replacement; Partial Arch Repair; Hemiarch Procedures; Total Arch Replacement (TARP); Frozen Elephant Trunk (FET) Hemiarch Procedures; Type B Acute Aortic Dissection (TBAAD); Type B non acuteAortic Dissection (TBAD)
MeSH Terms: conditions — Dissection, Ascending Aorta; Aortic Diseases; Aortic Valve Insufficiency | interventions — TARP; Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Ascending Aorta Replacement (AAR) with or without Hemiarch Repair: Patients who will require a conservative prosthetic replacement of the ascending aorta with or without hemiarch.Patients who required a concomitant aortic valve replacement with conventional xenograft or mechanical prosthesis
  Interventions: Procedure: Conservative Root- Sparing Aortic Valve Resuspension with or without Hemiarch Repair
- Ascending Aorta Replacement (AAR) with Aortic Root Replacement (ARR): Patient who will require the extensive procedure including ascending aorta replacement associated to root replacement with or without sparing of the aortic valve
  Interventions: Procedure: Extensive Ascending Aorta Replacement (AAR) with Aortic Root Replacement (ARR)
- Ascending Aorta Replacement with Total Arch Replacement (TARP): Patient who will require the extensive procedure including ascending aorta replacement associated to TARP
  Interventions: Procedure: Extensive Ascending Aorta Replacement (AAR) with Total Arch Replacement (TARP)
- Root and Ascending Aorta Replacement with Total Arch Replacement: Patient who will require the extensive procedure including root and ascending aorta replacement associated to TARP
  Interventions: Procedure: Extensive Root and Ascending Aorta Replacement with Total Arch Replacement
- Thoracic Endovascular Aortic Repair: Patient who will require the procedure including thoracic endovascular aorta repair
  Interventions: Procedure: Thoracic Endovascular Aortic Repair
- Open Thoracic Aortic Repair: Patient who will require the procedure including open thoracic aorta repair
  Interventions: Procedure: Open Thoracic Aortic Descendig Repair

INTERVENTIONS:
Procedure: Conservative Root- Sparing Aortic Valve Resuspension with or without Hemiarch Repair — Cardiac arrest will be performed by administering a potassium-rich antegrade cardioplegia solution delivered directly into the coronary ostium or in the case of aortic regurgitation after insertion of the coronary sinus cannula.The aorta will be resected up to the sinotubular junction and the thrombus located in the false lumen of the aortic root will be removed so that the aortic lesion can be visualized. The commissures will be resuspended using 4-0 or 5-0 sutures reinforced with a Teflon pledget above every commissure. A 4-0 or 5-0 polypropylene suture will be chosen to seal the proximal anastomosis and this suture line will also be used to secure the intima to the adventitia. In patients demonstrating normal-sized aortic roots associated with poor-quality valve leaflets, concomitant aortic valve replacement with conventional xenograft or mechanical prosthesis will be preferable.
  Other Names: Ascending Aorta Replacement with Aortic Valve Replacement (AVR)
  Groups: Ascending Aorta Replacement (AAR) with or without Hemiarch Repair
Procedure: Extensive Ascending Aorta Replacement (AAR) with Aortic Root Replacement (ARR) — Patients who experienced dilatation of the sinuses of Valsalva > 4.5 cm in diameter on computed tomography imaging, those with connective tissue disease, or those in whom intimal tears extended into the sinuses, will receive replacement of the aortic root using a biologic or mechanical composite valve graft or valve-sparing root reimplantation procedure associated to AAR
  Other Names: ARR with or without aortic valve sparing
  Groups: Ascending Aorta Replacement (AAR) with Aortic Root Replacement (ARR)
Procedure: Extensive Ascending Aorta Replacement (AAR) with Total Arch Replacement (TARP) — Total arch replacement procedures (TARP) will performed with the use of deep hypothermic circulatory arrest and with either antegrade or retrograde cerebral perfusion, maintaining systemic cooling between 19°C to 25°C and depending on the surgeon's practice.TARPs will be carried out using 1- and 4-branch grafts and involved the resection of all the aortic tissue up to the left common carotid artery (total arch)
  Other Names: AAR with TARP or Frozen Elephant Trunk (FET)
  Groups: Ascending Aorta Replacement with Total Arch Replacement (TARP)
Procedure: Extensive Root and Ascending Aorta Replacement with Total Arch Replacement — This extensive procedure will include complete replacement of the anterior thoracic aorta extending to part or all of the aortic arch. It will be performed with the previously reported techniques
  Other Names: Full anterior thoracic aorta replacement with partial hemiarch repair or TARP or FET
  Groups: Root and Ascending Aorta Replacement with Total Arch Replacement
Procedure: Thoracic Endovascular Aortic Repair — TEVAR patients have a higher incidence of complications and reintervention than open repair patients. TEVAR complications may include endoleak, retrograde type A aortic dissection, stent-graft migration, fracture or collapse, and increased size.
  Other Names: TEVAR
  Groups: Thoracic Endovascular Aortic Repair
Procedure: Open Thoracic Aortic Descendig Repair — Surveillance imaging can detect complications of open repair, such as graft infection and anastomotic pseudoaneurysm. After open repair or TEVAR, patients may develop progressive aneurysmal dilatation of adjacent or remote aortic segments.
  Other Names: TOAR
  Groups: Open Thoracic Aortic Repair

SUMMARY:
Type A aortic dissection (TAAD) is a potentially life-threatening pathology associated with significant risk of mortality and morbidity. In acute forms of type A aortic dissection (TAAD) mortality is 50% by 24 h and 50% of patients die before reaching a specialist center. Rapid diagnosis and subsequent prompt surgical repair remain the primary goal for these patients.

In the last decade it has been observed that improvements in diagnostic techniques, initial management and increased clinical awareness have contributed to a substantial increase in the number of patients benefiting from a prompt diagnosis and undergoing surgery.However, survival after surgical repair has not yet reached optimal follow-ups and is burdened by high in-hospital mortality(16-18%)The main approach to acute type B non-complicated aortic dissection (TBAD) has always been to use medicines to control the patient's heart rate and blood pressure. However, recent findings suggest that a large number of patients treated for acute complicated (TBAAD) and non-complicated TBAD experience aortic complications, such as aneurysmal degeneration, at a later stage.

DETAILED DESCRIPTION:
For patients requiring surgical repair for a TAAD, there is still some disagreement regarding which factors should be considered during the preoperative evaluation, the best decision-making process to undertake that best assesses procedural risk, and how operative mortality can be predicted. Furthermore, the impact of different surgical strategies on outcomes remains unclear.This prospective study was designed to evaluate the impact of the center volume-outcome relationship and that on mortality which remain poorly understood. A better understanding of the determinants of outcome in patients undergoing surgery could support decision making, aid in the design of service delivery, and improve outcomes for surviving patients who are referred to specialized centers for treatment of aortic disease.Furthermore, the study aims to evaluate whether precise risk stratification can provide better patient counseling and be used for unit-surgeon benchmarking. Ultimately in the present study, we aimed to investigate outcome predictors in patients undergoing surgery for TAAD, including clinical and perioperative variables as well as to evaluate follow up beyond 15 years.TBAD occurring beyond the left subclavian artery (LSA) is classified in chronological order based on the timing of clinical presentation: acute (14 days or less), subacute (more than 14 days and less than or equal to 3 months), and chronic (more than 3 months).TBADs are also divided into complicated or non-complicated based on their initial clinical manifestation. Acute complicated TBAD is characterised by tearing of the aorta, pain, rapid expansion, hypertension, or blockages in the vasculature.Malperfusion syndrome is the most common complication, occurring in nearly 30% of cases. More than 30% of patients with mesenteric compromise following aortic dissection die .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years
* TAAD or intramural hematoma involving the ascending aorta
* Symptoms started within 7 days from surgery
* Primary surgical repair of acute TAAD
* Any other major cardiac surgical procedure concomitant with surgery for TAAD.

Exclusion Criteria:

* Patients aged < 18 years
* Onset of symptoms > 7 days from surgery
* Prior procedure for TAAD
* Concomitant endocarditis;
* TAAD secondary to blunt or penetrating chest trauma.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The STAAD study is a prospective multicenter registry including patients who will underwent surgery for acute TAAD at 6 centers of cardiac surgery located in 2 European countries and Japan (3 France, 2 Italy and 1 Hokkaido ). Data will be prospectively collected from patients (conservative vs estensive Type A aortic dissection repair) who will be treated during the study period. In addition, the aim will be to gather further data for future clinical research on this topic. Preoperative and postoperative variables will be included during in-hospital stay and follow-up data instead they will be included on subsequent encounters for all other patients who will be hospitalized.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2005-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Operative Mortality (OM) | 30-day
  Patients who died within 30 days
Rate of mesenteric ischemia | 30-day
  Rate of abdominal pain with or without nausea and vomiting and rectal bleeding or bloody diarrhea
Rate of permanent Neurologic Deficit (PND) | 30-day
  Number of participants with acute episode of a focal or global neurological deficit. Rates of alteration of degree of consciousness, hemiplegia, hemiparesis, numbness or sensory loss affecting one side of the body, dysphasia or aphasia, hemianopsia, amaurosis fugax. To consider rate of other neurologic signs or symptoms consistent with stroke duration of focal or global neurologic deficit greater than 24 hours.
Rate of composite of Major Adverse Events (MAE) | 30-day
  Number of participants with MAE which will include the composite rate of myocardial infarction, cerebrovascular accident, need for dialysis, or need for tracheostomy according to Common Terminology Criteria for Adverse Events v4.0 (CTCAE)
Rate of perioperative Myocardial Infarction (MI) | 30-day
  Number of participants with MI based on fourth universal definition.
Rate of acute heart failure (AHF) | 30-day and in-hospital mortality
  Number of participants with postoperative AHF who will require prolonged use of concentration of inotropes for a period greater than 24 h and/or the insertion of any mechanical circulatory support device.

SECONDARY OUTCOMES:
Rate of Transient Neurologic Deficit (TND) | 30-day
  Number of participants who will complicate postoperatively with episode of TND which will include complication rate such as confusion, delirium, agitation
Rate of spinal Cord Injury (SCI) | 30-day
  Number of participants with SCI intended as rate of paraplegia and/or paraparesis
Rate of acute kidney injury | 30-day
  Number of participants with postoperative change in serum creatinine concentration. Severity will be stratified on the basis of number of participants with the KDIGO (Kney Disease Improving Global Outcomes) criteria.
Rate of perioperative bleeding | 30-day
  Number of participants who will receive postoperative transfused red blood cell units. The E-CABG ( coronary artery by pass grafting) classification of bleeding rate has been proposed as a simple classification of perioperative bleeding
Reoperation for bleeding | 30-day
  Number of participants who will receive postoperative chest reopening for excessive bleeding.
Rate of mechanical circulatory support | 30-day
  Number of participants who will receive the use of intra-aortic balloon pump and/or venoarterial extracorporeal membrane oxygenation for postoperative acute heart failure.
Rate of composite of Major Adverse Pulmonary Events (MAPE) | 30-day
  Number of participants with MAPE which will include the composite rate of intubation >48 hours, pneumonia, reintubation, tracheostomy according to the Common Terminology Criteria for Adverse Events v4.0 (CTCAE)
Rate of reintervention | 18-years
  The number of participants who will require reoperation for the aortic valve, proximal aorta, or distal aorta.
Rate of late survival | 18-years
  Data on patient's survival status will be collected

OTHER OUTCOMES:
Rate of urgent procedure | 30-day
  Number of participants who will require scheduled procedure within 24 hours of admission.
Rate of emergency grade 1 | 30-day
  Number of participants will require procedure within 24 hours of hospital admission and who are symptomatic or minimally symptomatic with stable hemodynamic conditions and no signs of malperfusion.
Rate of emergency grade 2 | 30-day
  Number of participants who will require procedure within the first 6 hours of hospital admission due to hemodynamic instability despite use of concentration inotropes and/or malperfusion.
Rate of salvage grade 1 | 30-day
  Number of participants who will require immediate surgical procedure. Rate of cardio pulmonary resuscitation with external chest compressions and/or open cardiac massage between induction of anesthesia and initiation of cardiopulmonary bypass.
Rate of salvage grade 2 | 30-day
  Number of participants who will require immediate surgical procedure. Rate of cardiopulmonary resuscitation with external chest compressions en route to the operating theatre or prior to induction of anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Nappi, MD, Study Chair — Cardiac Surgery Centre Cardiologique du Nord de Saint-Denis, Paris, France
Locations (1):
- Francesco Nappi, Saint-Denis, France

REFERENCES:
- [Result] Mahase E. Half of patients with acute aortic dissection in England die before reaching a specialist centre. BMJ. 2020 Jan 23;368:m304. doi: 10.1136/bmj.m304. No abstract available. PMID 31974270
- [Result] Braverman AC. Acute aortic dissection: clinician update. Circulation. 2010 Jul 13;122(2):184-8. doi: 10.1161/CIRCULATIONAHA.110.958975. No abstract available. PMID 20625143
- [Result] Howard DP, Banerjee A, Fairhead JF, Perkins J, Silver LE, Rothwell PM; Oxford Vascular Study. Population-based study of incidence and outcome of acute aortic dissection and premorbid risk factor control: 10-year results from the Oxford Vascular Study. Circulation. 2013 May 21;127(20):2031-7. doi: 10.1161/CIRCULATIONAHA.112.000483. Epub 2013 Apr 18. PMID 23599348
- [Result] Biancari F, Juvonen T, Fiore A, Perrotti A, Herve A, Touma J, Pettinari M, Peterss S, Buech J, Dell'Aquila AM, Wisniewski K, Rukosujew A, Demal T, Conradi L, Pol M, Kacer P, Onorati F, Rossetti C, Vendramin I, Piani D, Rinaldi M, Ferrante L, Quintana E, Pruna-Guillen R, Rodriguez Lega J, Pinto AG, Acharya M, El-Dean Z, Field M, Harky A, Nappi F, Gerelli S, Di Perna D, Gatti G, Mazzaro E, Rosato S, Raivio P, Jormalainen M, Mariscalco G. Current Outcome after Surgery for Type A Aortic Dissection. Ann Surg. 2023 Oct 1;278(4):e885-e892. doi: 10.1097/SLA.0000000000005840. Epub 2023 Mar 13. PMID 36912033
- [Result] Benedetto U, Dimagli A, Kaura A, Sinha S, Mariscalco G, Krasopoulos G, Moorjani N, Field M, Uday T, Kendal S, Cooper G, Uppal R, Bilal H, Mascaro J, Goodwin A, Angelini G, Tsang G, Akowuah E. Determinants of outcomes following surgery for type A acute aortic dissection: the UK National Adult Cardiac Surgical Audit. Eur Heart J. 2021 Dec 28;43(1):44-52. doi: 10.1093/eurheartj/ehab586. PMID 34468733
- [Result] Geirsson A, Shioda K, Olsson C, Ahlsson A, Gunn J, Hansson EC, Hjortdal V, Jeppsson A, Mennander A, Wickbom A, Zindovic I, Gudbjartsson T. Differential outcomes of open and clamp-on distal anastomosis techniques in acute type A aortic dissection. J Thorac Cardiovasc Surg. 2019 May;157(5):1750-1758. doi: 10.1016/j.jtcvs.2018.09.020. Epub 2018 Sep 29. PMID 30401530
- [Result] Harris KM, Nienaber CA, Peterson MD, Woznicki EM, Braverman AC, Trimarchi S, Myrmel T, Pyeritz R, Hutchison S, Strauss C, Ehrlich MP, Gleason TG, Korach A, Montgomery DG, Isselbacher EM, Eagle KA. Early Mortality in Type A Acute Aortic Dissection: Insights From the International Registry of Acute Aortic Dissection. JAMA Cardiol. 2022 Oct 1;7(10):1009-1015. doi: 10.1001/jamacardio.2022.2718. PMID 36001309
- [Result] Czerny M, Schoenhoff F, Etz C, Englberger L, Khaladj N, Zierer A, Weigang E, Hoffmann I, Blettner M, Carrel TP. The Impact of Pre-Operative Malperfusion on Outcome in Acute Type A Aortic Dissection: Results From the GERAADA Registry. J Am Coll Cardiol. 2015 Jun 23;65(24):2628-2635. doi: 10.1016/j.jacc.2015.04.030. PMID 26088302
- [Result] O'Hara D, McLarty A, Sun E, Itagaki S, Tannous H, Chu D, Egorova N, Chikwe J. Type-A Aortic Dissection and Cerebral Perfusion: The Society of Thoracic Surgeons Database Analysis. Ann Thorac Surg. 2020 Nov;110(5):1461-1467. doi: 10.1016/j.athoracsur.2020.04.144. Epub 2020 Jun 26. PMID 32599034